CLINICAL TRIAL: NCT02360033
Title: Systemic Therapy and Cognitive Behavioral Therapy for Social Anxiety Disorders With Adults: Manual Development and Randomized-Controled Feasibility Study
Brief Title: Systemic Therapy and Cognitive Behavioral Therapy for Social Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: German Association for Systemic Therapy, Counseling and Family Therapy (DGSF) (Unknown); Systemic Society (SG) (Unknown); Heidehof Foundation (Unknown)
Responsible Party: Principal Investigator, Christina Hunger, Principal Investigator, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOPHO-PT-2014
Record Dates: First submitted 2015-01-21; First posted 2015-02-10 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systemic Therapy (Experimental): Systemic Therapy deals with the experience in private social systems (e.g. couples. Family, friends) and organizational systems (e.g. work teams), their appraisals and the attitude of the members towards each other within the system. It is analyzed how these systems can lead to the development and maintenance of psychological disorders.
  Interventions: Behavioral: Systemic Therapy for Social Anxiety Disorder
- Cognitive Behavioral Therapy (Experimental): Cognitive Behavioral Therapy deals with individual behavior as well as individual attitude, thoughts, appraisals and beliefs, which can have an influence on the development and maintenance of psychological disorders.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Social Anxiety Disorder

INTERVENTIONS:
Behavioral: Systemic Therapy for Social Anxiety Disorder
  Arms: Systemic Therapy
Behavioral: Cognitive Behavioral Therapy for Social Anxiety Disorder
  Arms: Cognitive Behavioral Therapy

SUMMARY:
Goals of the study:

Systemic Therapy was approved in 2008 by the Scientific Advisory Board on Psychotherapy (Wissenschaftlicher Beirat Psychotherapie: WBP) for a variety of disorders which, at the time, did not include anxiety disorders. According to the 2007 joint methods paper of the WBP and the Mutual Federal Committee (Gemeinsamen Bundesausschuss: G-Ba), there must be three randomized-controlled trials (RCT) for anxiety disorders. These studies are available now but lack explicit details about the clinical significance of the reductions they show in social anxiety symptoms. This project is funded by the German Association for Systemic Therapy, Counseling and Family Therapy (Deutsche Gesellschaft für Systemische Therapie, Beratung und Familientherapie: DGSF).

Study design:

The study is planned as a mono-centric, balanced pilot RCT. It investigates the feasibility of an RCT comparing Systemic Therapy and Cognitive Behavioral Therapy for Social Anxiety Disorders (SAD) in 32 patients.

ELIGIBILITY:
Inclusion Criteria:

* Social Anxiety Disorder (SKID: ICD-Diagnosis: F40.1, Liebowitz Social Anxiety Scale > 30);
* Agreement to participate in the study and to be randomized into the two treatment groups

Exclusion Criteria:

* Acute drug or alcohol intoxication or dependency
* Anorexia with BMI < 14
* Psychotic disorder
* Severe physical diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change of Liebowitz Social Anxiety Scale (LSAS-SR) | Baseline, 8th,15th, 20th and 26th hour of therapy; 6, 9 and 12 months after randomization
  Social Anxiety will be assessed using the Liebowitz Social Anxiety Scale (LSAS-SR) in its German version. The LSAS-SR is a brief 24-item self report instrument with 13 items relating to performance anxiety and 11 concerning social situations. Its purpose is to assess the range of social interaction and performance situations feared and the degree of avoidance by a patient in order to assist in the diagnosis of social anxiety disorder, 24 items, German version
Change of Social Interaction Anxiety Scale (SIAS) | Baseline, 8th,15th, 20th and 26th hour of therapy; 6, 9 and 12 months after randomization
  Measure of social interaction anxiety, 20 items, German version
Change of Social Phobia Scale (SPS) | Baseline, 8th,15th and 20th hour of therapy, end of treatment; 6, 9 and 12 months after randomization
  Measure of anxiety while being observed by others, 20 items, German version

SECONDARY OUTCOMES:
Change of Adjustment to Symptomatology Scale (ASS) | Baseline, 8th,15th, 20th and 26th hour of therapy; 6, 9 and 12 months after randomization
  Measure of adjustment to the symptomatology, 5 items, German version
Change of Evaluation of Social Systems (EVOS) | Baseline, 8th,15th, 20th and 26th hour of therapy; 6, 9 and 12 months after randomization
  Measure of social relationships in different social systems, 10 items, German version
Change of Experience in Social Systems (EXIS) | Baseline, 8th,15th, 20th and 26th hour of therapy; 6, 9 and 12 months after randomization
  Measure of the individual experience in different social systems, 24 items, German version
Change of Beck Depression Inventory-II (BDI-II) | Baseline, 8th,15th, 20th and 26th hour of therapy; 6, 9 and 12 months after randomization
  Severity of depressive symptoms "at that moment", specifically assessing the intensity of depression in psychiatric and normal populations, 21 items, German version
Change of Brief Symptom Checklist (BSCL) | Baseline, 8th,15th, 20th and 26th hour of therapy; 6, 9 and 12 months after randomization
  The instrument provides an overview of a patient's symptoms and their intensity at a specific point in time, 53 items, German version
Change of Inventory of Interpersonal Problems (IIP-32) | Baseline, 8th,15th, 20th and 26th hour of therapy; 6, 9 and 12 months after randomization
  The IIP-32 is a self-report instrument that identifies a person's most salient interpersonal difficulties. It is a short version of the Inventory of Interpersonal Problems, 32 items, German version
Change of Dyadic Adjustment Scale (DAS-12) | Baseline, 8th,15th, 20th and 26th hour of therapy; 6, 9 and 12 months after randomization
  Measure of relationship adjustment, 12 items, German version
Change of University of Rhode Island Change Assessment (URICA-S, short version) | Baseline, 8th,15th, 20th and 26th hour of therapy; 6, 9 and 12 months after randomization
  Measure of stages of change, 16 items, German version
Change of Burden Assessment Scale (BAS) | Baseline, 26th hour of therapy; 12 months after randomization
  Measure of perceived burden in daily life among resource persons, 19 items, German version
Change of Scale for the Multiperspective Assessment of General Change Mechanisms in Psychotherapy (SACiP), | 8th,15th, 20th and 26th hour of therapy; 6, 9 and 12 months after randomization
  Measure of the six dimensions of resource activation, problem actuation, mastery, clarification of meaning, emotional bond, agreement on collaboration, 21 items, German version

CONTACTS AND LOCATIONS:
Overall Officials: Christina Hunger, Dr., Study Director — Institute of Medical Psychology, University Hospital Heidelberg/Germany; Jochen Schweitzer, Prof. Dr., Study Chair — Institute of Medical Psychology, University Hospital Heidelberg/Germany; Hinrich Bents, Dr., Study Chair — Centre for Psychological Psychotherapy Heidelberg (ZPP)
Locations (1):
- Institute of Medical Psychology, University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Hunger C, Hilzinger R, Koch T, Mander J, Sander A, Bents H, Schweitzer J. Comparing systemic therapy and cognitive behavioral therapy for social anxiety disorders: study protocol for a randomized controlled pilot trial. Trials. 2016 Mar 31;17:171. doi: 10.1186/s13063-016-1252-1. PMID 27029546
- See also: Related Info — https://www.klinikum.uni-heidelberg.de/